CLINICAL TRIAL: NCT02225496
Title: A Phase II Study of Transoral Robotic Surgery With Adjuvant Therapy for Surgically Resectable HPV-positive Oropharyngeal Cancer
Brief Title: Robotic Surgery for Oropharyngeal Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Another trial in the department directly competes for the the same patient population
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0925; NCI-2014-02126 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Oropharyngeal Cancer
Keywords: Oropharyngeal cancer; Oropharynx; Human papilloma virus; HPV positive; Squamous cell carcinoma; SCC; Transoral robotic surgery; TORS; Intuitive Surgical da Vinci Surgical System; Modified barium swallow; MBS; Questionnaires; Surveys; Speech and swallowing function
MeSH Terms: conditions — Oropharyngeal Neoplasms; Carcinoma, Squamous Cell; Speech | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transoral Robotic Surgery (TORS) (Experimental): Transoral robotic surgery performed utilizing Intuitive Surgical da Vinci Surgical System. Utilizing robotic surgical system, tumor excised with wide surgical margins of 0.5-1 cm. Functional assessment performed at pre-treatment, within 1-4 weeks post-op from TORS (before adjuvant therapy), and after completion of treatment at the following time points: 6 months (±2 months), 12 months (±2 months), and 24 months (±6 months). Functional measures include video-fluoroscopic examination of swallowing (modified barium swallow [MBS] study) with administration of the Performance Status Scale-Head and Neck (PSS-HN) and MD Anderson Dysphagia Inventory (MDADI) questionnaire.
  Interventions: Procedure: Transoral Robotic Surgery (TORS); Procedure: Modified Barium Swallow (MBS); Behavioral: Questionnaires

INTERVENTIONS:
Procedure: Transoral Robotic Surgery (TORS) — Transoral robotic surgery performed utilizing Intuitive Surgical da Vinci Surgical System. Utilizing robotic surgical system, tumor excised with wide surgical margins of 0.5-1 cm.
Procedure: Modified Barium Swallow (MBS) — MBS performed at baseline and 1 - 4 weeks after surgery, and at 6 months, 12 months and 24 months.
  Other Names: MBS
Behavioral: Questionnaires — Questionnaires about speech and swallowing function completed at baseline, 1 - 4 weeks after surgery, and at 6 months, 12 months, and at 24 months.
  Other Names: Surveys

SUMMARY:
Standard-of-care treatment options for oropharyngeal cancer often result in long-term side effects that interfere with normal quality of life. A minimally-invasive transoral robotic surgery (TORS) approach has been developed to operate on the disease site while affecting the surrounding tissue as little as possible. Researchers think that this approach may help to control the disease and avoid such long-term side effects.

The goal of this clinical research study is to learn if minimally-invasive transoral robotic surgery (TORS) can help to control HPV-positive oropharyngeal cancer. Transoral means through the mouth. The TORS approach is called the Intuitive Surgical da Vinci Surgical System.

Researchers also want to learn if this surgery affects participants' ability to speak and swallow.

DETAILED DESCRIPTION:
Study Surgery:

If you are found to be eligible to take part in this study, you will be scheduled for surgery. You will receive general anesthesia to make you sleep during the procedure. You will be asked to sign a separate consent form that describes the anesthesia and its risks. If the doctor thinks it is needed, the abnormal area will be looked at with a tube that has a lighted camera on one end (called a laryngoscopy) to check the size of the tumor and to look for any additional cancerous areas.

The tumor will be exposed with standard equipment after the teeth are protected with a dental guard. Using the robotic surgical system, the tumor will be removed.

Your affected lymph nodes will be surgically removed through your neck. The robotic system will not be used for that part of the surgery. The nerve that controls the shoulder, the blood vessel that brings blood back to the heart from the brain and neck, and the major muscle of the front of the neck will all be saved, unless the tumor in the lymph nodes has grown directly into those areas. A drain will be placed before the surgical wound is closed. The drain will usually be removed within a week after surgery.

Based on the results of surgery, you will receive adjuvant therapy (therapy after the surgery). For example, if your surgery does not remove enough of the cancer, you will be referred to receive radiation therapy. There will likely need to be a 1-2 week delay before you can receive radiation therapy. Your doctor will discuss this therapy with you in more detail, including the risks.

Length of Study:

The surgery will be stopped if the doctor thinks the tumor is too large to be removed with the robotic system. You will be taken off study if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits and data collection.

Follow-Up Visits:

Within 1-4 weeks after surgery (+/- 3 days):

* You will have a physical exam, including a cranial nerve exam of your tongue, palate, and facial nerves.
* You will have an MBS.
* You will meet with a speech pathologist.
* You will complete the questionnaires about your speech and swallowing function.

At 6 months (+/- 2 months), 12 months (+/- 2 months), and 24 months (+/- 6 months) after surgery:

* You will have an MBS.
* You will have a cranial nerve exam of your tongue, palate, and facial nerves.
* You will meet with a speech pathologist.
* You will complete the questionnaires about your speech and swallowing function.

As often as the doctor thinks it is needed for up to 5 years after surgery, the study staff will check your medical record to find out how you are doing and about any treatments and follow-up you have had.

This is an investigational study. The robotic surgical procedure (the daVinci Surgical System) is FDA approved and commercially available. The study doctor can explain how the surgery is designed to work.

Up to 150 participants will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a previously untreated, T1 or T2, N0-N2b transorally resectable (as determined by the treating surgeon), histologically proven HPV positive, squamous cell carcinoma (SCC) of the oropharynx.
2. Eastern Cooperative Oncology Group (ECOG) PS 0-2.
3. Age >/= 18 years.
4. Negative serum pregnancy test in females of childbearing potential.
5. Patients must sign a study-specific informed consent form prior to treatment.

Exclusion Criteria:

1. Evidence of distant metastases (below the clavicle) by clinical or radiographic examination.
2. Evidence of any other primary cancers or metastases. Evidence of deep soft-tissue or bony invasion, which would preclude TMIS by clinical and/or radiographic exam.
3. Contraindications to general anesthesia.
4. Patients who have had chemotherapy or radiotherapy to the oropharynx prior to entering the study.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
6. Patients with tumors whose resection would necessitate a free-tissue transfer for reconstruction of the surgical defect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Time to local-regional recurrence (TTLRR) | 6 months after surgery
  Primary efficacy endpoint is time to local-regional recurrence (TTLRR). TTLRR measured from surgery (using minimally-invasive Transoral Robotic Surgery (TORS)) date to first date that local-regional recurrence disease is objectively documented or to last follow-up date if local-regional recurrence has not occurred during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Kupferman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org